In the study of dry eye disease, it is being investigated whether symptoms of dry eye disease improve with the related treatment. Participation in this work will depend on the willingness of the volunteer, and voluntary withdrawal can be done without refusing to participate in the investigation without losing any right without any obligation. Treatment of dry eyes with 0.05% cyclosporine emulsion and artificial tears with 50% diluted autologous serum on dry eye symptoms was performed by using self-administered serum and eye drops to treat restasis tear drop and refresh artificial tear drip treatments individually I am committed to using the treatment as a combined treatment, completing the treatment protocol for 60 days, and filling the questionnaire for control surveys to respond to treatment. In case of any difficulties during the treatment, doctor. I give my consent to observational work for treatment purposes within the scope of my own request and provision, knowing that I will be able to reach by telephone and abandon the treatment in case of side effects.

Under these circumstances I have read all the explanations on the "Informed Volunteer Form". The written and oral explanations about the research mentioned above and aimed at me were made by the physician mentioned below. I know when I voluntarily participate in the research, I can leave without seeking justified or unjustified whenever I want "

Name / surname / signature / date of the volunteer Name / surname / signature / date of the researcher